CLINICAL TRIAL: NCT07244523
Title: Prospective, Comparative, Two-arms, Randomized, Controlled, Investigator/Assessor-blinded Study for the Evaluation of the Efficacy and Safety of a Medical Device With a Physical Mode of Action (X92001919) Versus Paranic Anti-lice Shampoo on the Treatment of Head Lice Infestation.
Brief Title: Efficacy and Safetyof a Medical Device With a Physical Mode of Action (X92001919) Versus Paranix Anti-lice Shampoo.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OYS013-0025
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lice; Head Lice
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, two-arms, randomized, controlled, investigator/assesor-blinded study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulverize (X92001919) (Experimental): Treatment with product Pulverize at Visit 1 (Day 0),Visit 2 (Day 3) and Visit 3 (Day 7). Counting alive lice and nymphs in the hair at Visit 1 (Day 0), Visit 2 (Day 3), Visit 3 (Day 7) and Visit 4 (Day 10).
  Interventions: Device: Pulverize (X92001919)
- Paranix Anti-Lice Shampoo (Active Comparator): Treatment with product Paranix Anti-Lice Shampoo at Visit 1 (Day 0) and Visit 3 (Day 7). Counting alive lice and nymphs in the hair at Visit 1 (Day 0), Visit 2 (Day 3), Visit 3 (Day 7) and Visit 4 (Day 10).
  Interventions: Device: Paranix Anti-Lice Shampoo

INTERVENTIONS:
Device: Pulverize (X92001919) — Treatment at Day 0, Day 3 and Day 7 with the Pulverize Dry Shampoo formulation (X92001919)
  Arms: Pulverize (X92001919)
Device: Paranix Anti-Lice Shampoo — Treatment at Day 0 and Day 7 with the Paranix Anti-Lice Shampoo
  Arms: Paranix Anti-Lice Shampoo

SUMMARY:
Comparison of the efficacy of a new medical device with a physical mode of action to Paranix anti-lice shampoo in the treatment of head lice infestation.

DETAILED DESCRIPTION:
Pediculosis capitis or head lice infestation is a human medical condition caused by the infestation of the hair by the parasitic insect Pediculus humanus capitis (human head lice). When lice feed, they inject saliva into the scalp. The saliva is an anticoagulant which keeps blood from clotting making their feeding process easier. Many individuals experience an allergic reaction to the saliva, causing up to 50% of the population with head lice to itch. For this reason, the most common symptom of infestation is pruritus (itching) on the head. The bite reaction is very mild and it can be rarely seen between the hairs. In rare cases, the itch scratch cycle can lead to secondary infection. Swelling of the local lymph nodes and fever are rare.

There are a range of interventions available for the management of head lice. The main stay of therapy has been largely dependent on insecticidal-based approaches for several decades. However, the accumulating evidence with resistance to frontline insecticidal treatments like pyrethrins, permethrin and malathion has led to a growing incentive to develop newer and more effective treatments to treat the condition safely [3]. Over the past couple of decades, alternative candidates have been introduced into the market, including products with a physical mode of action that works via dehydration and suffocation of the lice [4-8].

The tested product has been developed with the ambition to offer a complete and safe head lice treatment, highly effective against head lice and eggs, whilst also offering ultimate convenience in use - making treatment of head lice infestation easy, and effective in few minutes. This is a medical device, not yet on the market, with a physical mode of action of suffocation and dehydration. The comparator product, Paranix® Anti-Lice Shampoo, is a reference product with a physical mode of action, available on the market in Europe as a class I medical device.

The main objective of the current study is to evaluate the efficacy and safety on head lice treatment of the device X92001919 versus Paranix® Anti-Lice Shampoo comparator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (except head lice infestation) based on medical history;
* Gender: male or female;
* Age: 2 years and above at the time of enrolment ;
* Subject with a slight to moderate lice infestation (according to EU norms)
* Subjects with various hair type (from 1 to 3C in the hair scale below) and hair length (from short to mid length hair, not exceeding shoulder)
* Documented oral informed consent for all subjects, including minors, given freely and expressly before the start of the study
* Written informed consent for subjects ≥18 years or legal guardian for subjects < 18 years given freely and expressly before start of the study;
* Written assent for subjects ≥12 to <18 years.
* Subject/Subject's legal guardian is psychologically able to understand the study related information and to give written informed consent;
* Females of childbearing potential must have a negative pregnancy test before the beginning of the study and agree to use a reliable method of birth control during the study.
* Subject agrees not to cut or chemically treat their hair while participating in the study.
* Subjects agrees not to use any other anti-lice treatment or medicated hair grooming products for the duration of the study.

Exclusion Criteria:

* In terms of population

  1. Pregnant (confirmed by pregnancy test at D0 for women of childbearing potential) or nursing woman or planning a pregnancy during the study;
  2. Subject who had been deprived of their freedom by administrative or legal decision or adult subject who is under guardianship;
  3. Subject in a social or sanitary establishment;
  4. Subject in an exclusion period from a previous study or who is currently participating in another study on hair/scalp or who participated to another clinical study on hair/scalp within 3 months before first visit.
  5. Subject suspected to be non-compliant according to the Investigator's judgment.
  6. Subject with curly or frizzy hair (from 4A to 4C in the hair type scale above).
  7. Subject with hair length below the shoulder.
  8. Subjects with more than 24 lice on the head.
* In terms of associated pathology 9. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.

  10. Subject with a cutaneous disease on the studied zone (scalp and hair). 11. Subject with severe scratches or open wounds/skin damages on the scalp (lice bites allowed however).

  12. Subject with a known or suspected allergy to any of the components/materials of the investigational products, anti-lice comb or post- treatment shampoo.

  13. Subject who has diabetes (type 1 or 2). 14. Subject with known or suspected immune deficiency or autoimmune disease.
* Relating to previous or ongoing treatment 15. Subject undergoing a topical treatment on the test area or a systemic treatment with:

  * anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the study;
  * corticosteroids during the 2 previous weeks and during the study;
  * retinoids and/or immunosuppressors during the 3 previous months and during the study;
  * any medication stabilized for less than one month. 16. Subject who received an anti-lice treatment in the previous 2 months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Pulverize (X92001919) compared to the comparator Paranix Anti-Lice Shampo. | 10 days
  Evaluate the efficacy of Pulverize (X92001919) compared to the comparator Paranix Anti-Lice Shampoo on the treatment of head lice infestation, after one treatment consisting of 3 applications. Efficacy of the treatment will be defined as the cure rate at the end of day 10, corrected for re-infestation.

SECONDARY OUTCOMES:
Efficacy comparison (uncorrected for re-infestation) | 10 days
  Evaluate and compare the efficacy for both products. (cure rate at the end of day 10, uncorrected for re-infestation).
Cure rate on day 3 and day 7 | day 3 for cure rate of first application day 7/day 10 for second application (depending on treatment).
  Evaluation of the cure rate on day 3 and day 7 in both separate groups, and comparison of both product effect after only one (on day 3) or two applications (day 7 for Pulverize versus day 10 for Paranix).
Indirect efficacy on eggs and evaluate potential re-infestation | Treatment time (day 0 - day 10
  Presence of live lice and nymphs, for both groups and between groups, without combing on hair and close to scalp on day 0 (prior to treatment to assess severity of the infestation), day 3, day 7, and day 10.
  These evaluations will assess indirect efficacy on eggs and evaluate potential re-infestation.
General well-being of subject (Esthetical effect) | Day 0 and day 7 of the study
  Analysis of subject's (or subject's parents/guardians) questionnaire at day 0 and day 7 to evaluate esthetical effect of the product. A comparison of the answers will be performed between the two products.
Safety by Adverse Events (AEs) | Duration of the study (day 0 - day 10)
  Number and evaluation of Adverse Events (AEs) reported during the study.
Local tolerability on 5-point scales | Duration of study (day 0- day 10)
  For both products, evaluation of local tolerability by the dermatologist on 5-point scales including dandruff state, greasy scalp, erythema, desquamation dryness, burning sensation, paraesthesia and pruritus and on 4 point-scales including skin irritation and eye irritation, on D0 (before and after product application), D3 (before and after application), D7 (before and after product application) and D10.
Global tolerability | Day 10
  For both products, assessment of global tolerability by the dermatologist on day 10 on a 4-point scale.

IPD SHARING:
Plan to Share IPD: No